CLINICAL TRIAL: NCT01994538
Title: Seven Versus Fourteen Day Treatment for Male Urinary Tract Infection
Brief Title: Seven vs. 14 Days Treatment for Male Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-008-13S; I01BX007080 (Other Grant/Funding Number: VA Merit Review)
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Tract Infections; Urinary antiinfective agents
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Longer (14 day) duration antimicrobial treatment (Active Comparator): 14 days of ciprofloxacin or trimethoprim/sulfamethoxazole
  Interventions: Other: Longer therapy duration
- Shorter (7 day) duration antimicrobial treatment (Placebo Comparator): 7 days of ciprofloxacin or trimethoprim/sulfamethoxazole, followed by 7 days of placebo
  Interventions: Other: Shorter therapy duration

INTERVENTIONS:
Other: Longer therapy duration — 14 days of antimicrobial treatment
  Arms: Longer (14 day) duration antimicrobial treatment
Other: Shorter therapy duration — 7 days of antimicrobial treatment
  Arms: Shorter (7 day) duration antimicrobial treatment

SUMMARY:
This study will investigate the treatment of urinary tract infection in men. Specifically, the investigators are looking to see if shorter duration of antibiotics (7 days) is any worse than longer duration of antibiotics (14 days). The investigators will also study whether longer treatment leads to an increase in antibiotic resistant bacteria in the large intestine (colon), or an increase in drug side effects.

DETAILED DESCRIPTION:
The proposed study is a randomized placebo-controlled trial of treatment duration for male urinary tract infection (UTI). Specifically, 319 men with a UTI will be randomized to 7 vs. 14 days of antimicrobial treatment. The primary outcome is resolution of UTI symptoms, assessed 14 days after completing active antimicrobial treatment. Secondary outcomes include recurrent UTI in the 4 weeks after treatment, adverse drug events, and intestinal carriage of antimicrobial resistant Gram-negative bacilli. Subjects will be enrolled from the Primary Care Clinic and Emergency Department at the Minneapolis VA Medical Center (MVAMC).

Currently, the optimal treatment duration for male UTI is unknown. A clinical trial of 14 vs. 28 days of treatment showed no difference in outcomes, whereas another trial of 3 vs.14 days showed an increase in recurrence with 3 days of treatment. However, current treatment recommendations are to treat men with UTI for 7 to 14 days, and no data exist to favor the shorter or longer duration. Most men with UTI in the VA are treated for more than 7 days, which is associated with a small but significant increase in Clostridium difficile infection. Additionally, other studies of non-UTI infectious diseases have shown that longer-duration treatment leads to increased antimicrobial resistance. Longer-duration treatment is also more costly and inconvenient to patients. Thus, since longer-duration treatment is associated with some adverse outcomes, in order to justify longer-duration treatment thee must be some clinically significant benefit to the extended treatment.

Accordingly, the proposed randomized placebo-controlled trial of 319 men with UTI will test the hypothesis that 7 days of antimicrobial treatment is non-inferior for the resolution of UTI symptoms when compared to 14 days of treatment. This study will provide valuable information to VA patients and clinicians regarding a common and understudied clinical decision.

ELIGIBILITY:
Inclusion Criteria:

Must have all

* Male gender
* New-onset (within 7 days) of at least one of the following symptoms/findings: dysuria, urinary frequency, urgency, hematuria, perineal pain, supra-pubic pain, costovertebral angle tenderness, or flank pain
* Treated as an outpatient (Primary Care Center or Emergency Department), with < 24 hours observation in the hospital or Emergency Department following the time of initial diagnosis
* Prescribed treatment with at least 7 days, but not more than 14 days, of either ciprofloxacin or TMP-SMZ

Exclusion Criteria:

Must have none

* Admission to the hospital (for > 24h) at the time of diagnosis
* Documented fever at time of initial evaluation ( 38.0 Celsius)
* Previous enrollment in the study
* Treatment for UTI in past 14 days
* Not able to give informed consent
* Unwilling to return for study visit
* Symptoms thought more likely to be caused by a non-UTI diagnosis (e.g., urinary calculus, sexually transmitted infection, etc.)
* Other antimicrobial therapy (new or ongoing) prescribed for a non-UTI diagnosis (e.g., cellulitis, pneumonia, etc.)
* Treatment initiated with an empiric antimicrobial to which the organism isolated in the urine culture is non-susceptible based on standard laboratory criteria
* Treatment initiated with an empiric antimicrobial regimen that is underdosed, based on current guidelines and reviews

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study of UTI in men
Enrollment: 273 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri M Drekonja, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
No formal plan submitted at time of grant. Will handle such requests on a case-by-case basis with input from local privacy officer and institutional review board.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Anticipate will share data for 2 years after publication of the primary result manuscript
Access Criteria: Requests will be handled on a case-by-case basis with input from the local privacy officer and IRB.

REFERENCES:
- [Derived] Drekonja DM, Trautner B, Amundson C, Kuskowski M, Johnson JR. Effect of 7 vs 14 Days of Antibiotic Therapy on Resolution of Symptoms Among Afebrile Men With Urinary Tract Infection: A Randomized Clinical Trial. JAMA. 2021 Jul 27;326(4):324-331. doi: 10.1001/jama.2021.9899. PMID 34313686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled subjects are afebrile men with symptomatic urinary tract infection who were initially treated with 7-14 days of trimethoprim/sulfamethoxazole (TMP/SMZ) or ciprofloxacin by the treating clinician. Subjects were randomized prior to day 8 of treatment to an additional 7 days of their original study drug (14d group) or placebo (7d group.
Pre-assignment Details: Primary analysis was per-protocol, and included all subjects who took at least 26 of 28 doses of medication.
  Intention to treat analysis includes all randomized subjects.
Period: Overall Study
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
Started (One subject consented but was not randomized due to a miscommunication with the research pharmacy) | 136 | 136
Completed (A second site (Houston VA) was added mid-study, and began enrolling 1/2018) | 136 | 136
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (11.6) | 67.8 (11.6) | 67.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 136 | 136 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 126 | 127 | 253
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 26 | 49
  White | 105 | 107 | 212
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 136 | 136 | 272
Indwelling catheter use [Count of Participants; unit: Participants] | 8 | 8 | 16
Intermittent catheter use [Count of Participants; unit: Participants] | 23 | 24 | 47
Diabetes [Count of Participants; unit: Participants] | 60 | 46 | 106
CKD [Count of Participants; unit: Participants] | 14 | 8 | 22
Cerebrovascular accident [Count of Participants; unit: Participants] | 5 | 13 | 18
Spinal cord injury [Count of Participants; unit: Participants] | 6 | 5 | 11
HIV [Count of Participants; unit: Participants] | 2 | 2 | 4
Prostatic hypertrophy [Count of Participants; unit: Participants] | 47 | 56 | 103
Prostatitis [Count of Participants; unit: Participants] | 18 | 16 | 34
Prostate Cancer [Count of Participants; unit: Participants] | 23 | 21 | 44
Prior UTI [Count of Participants; unit: Participants] | 78 | 84 | 162
Incontinence [Count of Participants; unit: Participants] | 52 | 44 | 96
Urethral stricture [Count of Participants; unit: Participants] | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Resolution of UTI Symptoms 14 Days After Completing Active Antimicrobial Therapy
Description: This outcome will be assessed in a binary manner. Subjects with persistent UTI symptoms or having received further antimicrobials because of UTI symptoms will be considered to have not met the primary outcome, whereas those without persistent UTI symptoms and not having received further antimicrobials will be considered to have met the primary outcome.
Time Frame: 14 days
Population: Per-protocol analysis (including all subjects who took medication as directed, defined as at least 26 of 28 doses, missing no more than 2 consecutive doses)
Measure: Count of Participants; unit: Participants
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
Number analyzed (Participants) | 123 | 131
Participants | 111 | 122

2. Secondary Outcome: Recurrent UTI Within 28 Days of Completing Active Study Medication
Description: New onset of symptomatic UTI within the 28 day follow-up period
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
Number analyzed (Participants) | 123 | 131
Participants | 15 | 13

3. Secondary Outcome: Adverse Drug Event in the 28 Days After Completing Study Medication
Description: The incidence of adverse drug events, including nausea, vomiting, diarrhea, dizziness, headache, drug allergy, and C. difficile infection, both individually and in aggregate, will be compared between treatment groups
  This outcome is number of subjects experiencing ANY adverse drug event
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
Number analyzed (Participants) | 136 | 136
Participants | 29 | 26

4. Secondary Outcome: Intestinal Carriage of Antimicrobial-resistant Gram Negative Bacilli
Description: Intestinal carriage of antimicrobial-resistant Gram-negative bacilli after completing study medication, as compared to a baseline sample taken early in treatment. Antimicrobial resistance for this measure was defined as newly detected resistance to either of the study drugs, ciprofloxacin or trimethoprim/sulfamethoxazole.
Time Frame: 7 days
Population: of the 163 subjects who participated in the optional intestinal carriage sub-study, 65 had growth in both of the submitted stool samples and are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
Number analyzed (Participants) | 29 | 36
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Longer (14 Day) Duration Antimicrobial Treatment | Shorter (7 Day) Duration Antimicrobial Treatment
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/136
Other Adverse Events (participants affected / at risk) | 33/136 | 28/136
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Longer (14 Day) Duration Antimicrobial Treatment (N=136) | Shorter (7 Day) Duration Antimicrobial Treatment (N=136)
Any adverse event (General disorders) | 33 (51) | 28 (40) — Adverse events assessed were: C difficile, nausea, vomiting, diarrhea, dizziness, headache, allergic reaction, thrush, muscle/joint aches, abnormal blood sugars, and changes in warfarin dosing. Subjects may have more than one adverse event.

LIMITATIONS AND CAVEATS:
Goal enrollment was 290; actual enrollment of 273 slightly reduces power to detect minimally clinically significant difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT01994538/Prot_SAP_000.pdf